CLINICAL TRIAL: NCT01148719
Title: Triage of Reduced Exercise Tolerance in Frail Elderly
Acronym: TREE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, F.H. Rutten, Dr, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 311040302; NL30278.041.10 (Other: Medical ethics committee of the University Medical Center Utrecht); NTR2336 (Registry Identifier: Nederlands Trial Register)
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Heart Failure; Chronic Obstructive Pulmonary Disease
Keywords: Heart Failure; Chronic Obstructive Pulmonary Disease; Dyspnea; Elderly; Diagnosis; Primary health care
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Dyspnea; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Index group (Active Comparator): Patients in the index group receive the diagnostic triage instrument. This includes echocardiographic, electrocardiographic and spirometric measurements and blood testing.
  Interventions: Other: Index group
- Control (No Intervention): Participants receive care as usual.

INTERVENTIONS:
Other: Index group — Diagnostic triage strategy includes; electrocardiography, echocardiography, spirometry and blood testing
  Other Names: Diagnostic triage strategy
  Arms: Index group

SUMMARY:
Background of the study:

Many elderly suffer from reduced exercise tolerance or exercise induced shortness of breath (dyspnoea) which causes decreased mobility and restrictions in physical, psychological and social functioning. Patients commonly attribute this symptom to their age, and simply adjust their life style to it. Reduced exercise tolerance/dyspnoea is very common with prevalence rate of 20-60% of those aged 65 years and over. The main causus in the elderly are heart failure and chronic obstructive pulmonary disease (COPD). Both diseases have a high negative impact on the quality of life and are associated with frequent hospital admissions. Over-diagnosis, but more often under-diagnosis of heart failure and COPD is rather common in primary care. Establishing a diagnosis early in the course of the disease is useful because both diseases can be adequately and evidence-based treated. Therefore, an easy diagnostic triage-strategy followed bij direct treatment would be of great importance to asses and treat heart failure and COPD in elderly patient with shortness of breath.

Objective of the study:

Quantify how many frail elderly aged over 65 years with reduced exercise tolerance and/or exercise induced dyspnoea have previously unrecognised COPD and heart failure. Quantify the difference in prevalence of unrecognised COPD and heart failure between those who underwent the diagnostic triage compared to those who received care as usual. Quantify the effect of the diagnostic triage plus the additionally treatment changes on functionality and quality of life after 6 months compared to those who received care as usual. Quantify the cost-effectiveness of the diagnostic triage strategy compared to care as usual

Study design:

A clustered randomized diagnostic (follow-up) study

Study population:

First, pre-selection of patients aged over 65 years from 50 general practices is based on frailty. Frailty is based on the next criteria: use 5 or more different types of medical drugs chronically in the last year and/or have 3 or more chronic or vitality treating diseases (such as diabetes mellitus, COPD, heart failure, impaired vision). This will be done from the electronic medical files of the general practices. These elderly will receive the MRC questionnaire of dyspnoea and three additional questions related tot exercise intolerance. Those with any dyspnoea and/or reduced exercise tolerance will be invited to participate, except those with established heart failure and COPD.

Study parameters/outcome of the study:

Prevalence of latent heart failure and COPD. Difference in prevalence of latent heart failure and COPD between both groups.

Differences in functionality and quality of life after 6 months between both groups. Cost-effectiveness and experienced patient burden of the diagnostic triage strategy.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 65 years and older
* must have a minimum of three chronic or vitality threatening diseases and/or use five or more medical drugs chronically in the last year
* must have dyspnea and/or reduced exercise tolerance (scored by two short questionnaires)

Exclusion Criteria:

* patients with both confirmed COPD and heart failure (Spirometry performed < 1 year ago and heart failure confirmed by echocardiography)
* patients unable or unwilling to sign informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 841 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of latent heart failure and COPD. | 6 months
  Prevalence of latent heart failure and COPD. The prevalence in the index-group is calculated after all investigations are done. The prevalence in de control-group is derived from the electronical medical files of the general practitioner after a follow-up period of six months.

SECONDARY OUTCOMES:
Effectiveness of the diagnostic triage strategy | 6 months
  (Cost-)effectiveness of the diagnostic triage strategy.
Difference in prevalence of latent heart failure and COPD between both groups | 6 months
  Difference in prevalence of latent heart failure and COPD between both groups. The prevalence in index-group is calculated after all investigations are done. The prevalence in de control-group is derived from the electronical medical files of the general practitioner after a follow-up period of six months.

CONTACTS AND LOCATIONS:
Overall Officials: Frans H Rutten, Dr., Principal Investigator — UMC Utrecht
Locations (1):
- General practionners " de Grebbe", Rhenen, Netherlands

REFERENCES:
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] Mulrow CD, Lucey CR, Farnett LE. Discriminating causes of dyspnea through clinical examination. J Gen Intern Med. 1993 Jul;8(7):383-92. doi: 10.1007/BF02600079. No abstract available. PMID 8410400
- [Background] Landahl S, Steen B, Svanborg A. Dyspnea in 70-year-old people. Acta Med Scand. 1980;207(3):225-30. doi: 10.1111/j.0954-6820.1980.tb09710.x. PMID 7368988
- [Background] Hogg K, Swedberg K, McMurray J. Heart failure with preserved left ventricular systolic function; epidemiology, clinical characteristics, and prognosis. J Am Coll Cardiol. 2004 Feb 4;43(3):317-27. doi: 10.1016/j.jacc.2003.07.046. PMID 15013109
- [Background] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Background] Rutten FH, Cramer MJ, Grobbee DE, Sachs AP, Kirkels JH, Lammers JW, Hoes AW. Unrecognized heart failure in elderly patients with stable chronic obstructive pulmonary disease. Eur Heart J. 2005 Sep;26(18):1887-94. doi: 10.1093/eurheartj/ehi291. Epub 2005 Apr 28. PMID 15860516
- [Background] Swedberg K, Cleland J, Dargie H, Drexler H, Follath F, Komajda M, Tavazzi L, Smiseth OA, Gavazzi A, Haverich A, Hoes A, Jaarsma T, Korewicki J, Levy S, Linde C, Lopez-Sendon JL, Nieminen MS, Pierard L, Remme WJ; Task Force for the Diagnosis and Treatment of Chronic Heart Failure of the European Society of Cardiology. Guidelines for the diagnosis and treatment of chronic heart failure: executive summary (update 2005): The Task Force for the Diagnosis and Treatment of Chronic Heart Failure of the European Society of Cardiology. Eur Heart J. 2005 Jun;26(11):1115-40. doi: 10.1093/eurheartj/ehi204. Epub 2005 May 18. No abstract available. PMID 15901669
- [Background] Rutten FH, Cramer MJ, Lammers JW, Grobbee DE, Hoes AW. Heart failure and chronic obstructive pulmonary disease: An ignored combination? Eur J Heart Fail. 2006 Nov;8(7):706-11. doi: 10.1016/j.ejheart.2006.01.010. Epub 2006 Mar 13. PMID 16531114
- [Background] Remes J, Miettinen H, Reunanen A, Pyorala K. Validity of clinical diagnosis of heart failure in primary health care. Eur Heart J. 1991 Mar;12(3):315-21. doi: 10.1093/oxfordjournals.eurheartj.a059896. PMID 2040313
- [Background] Bednarek M, Maciejewski J, Wozniak M, Kuca P, Zielinski J. Prevalence, severity and underdiagnosis of COPD in the primary care setting. Thorax. 2008 May;63(5):402-7. doi: 10.1136/thx.2007.085456. Epub 2008 Jan 30. PMID 18234906
- [Background] Wheeldon NM, MacDonald TM, Flucker CJ, McKendrick AD, McDevitt DG, Struthers AD. Echocardiography in chronic heart failure in the community. Q J Med. 1993 Jan;86(1):17-23. PMID 8438044
- [Background] Geijer RM, Sachs AP, Hoes AW, Salome PL, Lammers JW, Verheij TJ. Prevalence of undetected persistent airflow obstruction in male smokers 40-65 years old. Fam Pract. 2005 Oct;22(5):485-9. doi: 10.1093/fampra/cmi049. Epub 2005 Jun 17. PMID 15964866
- [Background] Rutten FH, Moons KG, Cramer MJ, Grobbee DE, Zuithoff NP, Lammers JW, Hoes AW. Recognising heart failure in elderly patients with stable chronic obstructive pulmonary disease in primary care: cross sectional diagnostic study. BMJ. 2005 Dec 10;331(7529):1379. doi: 10.1136/bmj.38664.661181.55. Epub 2005 Dec 1. PMID 16321994
- [Background] McHorney CA, Ware JE Jr, Raczek AE. The MOS 36-Item Short-Form Health Survey (SF-36): II. Psychometric and clinical tests of validity in measuring physical and mental health constructs. Med Care. 1993 Mar;31(3):247-63. doi: 10.1097/00005650-199303000-00006. PMID 8450681
- [Background] Aaronson NK, Muller M, Cohen PD, Essink-Bot ML, Fekkes M, Sanderman R, Sprangers MA, te Velde A, Verrips E. Translation, validation, and norming of the Dutch language version of the SF-36 Health Survey in community and chronic disease populations. J Clin Epidemiol. 1998 Nov;51(11):1055-68. doi: 10.1016/s0895-4356(98)00097-3. PMID 9817123
- [Background] Brooks RG, Jendteg S, Lindgren B, Persson U, Bjork S. EuroQol: health-related quality of life measurement. Results of the Swedish questionnaire exercise. Health Policy. 1991 Jun;18(1):37-48. doi: 10.1016/0168-8510(91)90142-k. PMID 10112300
- [Background] Weinberger M, Samsa GP, Schmader K, Greenberg SM, Carr DB, Wildman DS. Comparing proxy and patients' perceptions of patients' functional status: results from an outpatient geriatric clinic. J Am Geriatr Soc. 1992 Jun;40(6):585-8. doi: 10.1111/j.1532-5415.1992.tb02107.x. PMID 1587975
- [Background] Weber M, Hamm C. Role of B-type natriuretic peptide (BNP) and NT-proBNP in clinical routine. Heart. 2006 Jun;92(6):843-9. doi: 10.1136/hrt.2005.071233. No abstract available. PMID 16698841
- [Background] Wright SP, Doughty RN, Pearl A, Gamble GD, Whalley GA, Walsh HJ, Gordon G, Bagg W, Oxenham H, Yandle T, Richards M, Sharpe N. Plasma amino-terminal pro-brain natriuretic peptide and accuracy of heart-failure diagnosis in primary care: a randomized, controlled trial. J Am Coll Cardiol. 2003 Nov 19;42(10):1793-800. doi: 10.1016/j.jacc.2003.05.011. PMID 14642690
- [Background] Doust JA, Glasziou PP, Pietrzak E, Dobson AJ. A systematic review of the diagnostic accuracy of natriuretic peptides for heart failure. Arch Intern Med. 2004 Oct 11;164(18):1978-84. doi: 10.1001/archinte.164.18.1978. PMID 15477431
- [Background] Davie AP, Francis CM, Love MP, Caruana L, Starkey IR, Shaw TR, Sutherland GR, McMurray JJ. Value of the electrocardiogram in identifying heart failure due to left ventricular systolic dysfunction. BMJ. 1996 Jan 27;312(7025):222. doi: 10.1136/bmj.312.7025.222. No abstract available. PMID 8563589
- [Derived] van Mourik Y, Rutten FH, Bertens LCM, Cramer MJM, Lammers JJ, Gohar A, Reitsma JB, Moons KGM, Hoes AW. Clinical research study implementation of case-finding strategies for heart failure and chronic obstructive pulmonary disease in the elderly with reduced exercise tolerance or dyspnea: A cluster randomized trial. Am Heart J. 2020 Feb;220:73-81. doi: 10.1016/j.ahj.2019.08.021. Epub 2019 Sep 1. PMID 31790904
- [Derived] Bertens LC, Reitsma JB, van Mourik Y, Lammers JW, Moons KG, Hoes AW, Rutten FH. COPD detected with screening: impact on patient management and prognosis. Eur Respir J. 2014 Dec;44(6):1571-8. doi: 10.1183/09031936.00074614. Epub 2014 Jun 12. PMID 24925924
- [Derived] van Mourik Y, Moons KG, Bertens LC, Reitsma JB, Hoes AW, Rutten FH. Triage of frail elderly with reduced exercise tolerance in primary care (TREE). A clustered randomized diagnostic study. BMC Public Health. 2012 May 28;12:385. doi: 10.1186/1471-2458-12-385. PMID 22640176
- See also: study protocol — http://www.biomedcentral.com/1471-2458/12/385